CLINICAL TRIAL: NCT06648044
Title: Research of Therapeutic Targets in the Frame of Nephronophthisis and Renal Associated Ciliopathies - NPH_1
Brief Title: Research of Therapeutic Targets in the Frame of Nephronophthisis and Renal Associated Ciliopathies
Acronym: NPH1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMIS2015-05
Record Dates: First submitted 2024-01-23; First posted 2024-10-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Nephronophthisis; NPH1; Autosomal; Recessive; Genetically; Heterogenic; Disorder
Keywords: mutations; 20; genes
MeSH Terms: conditions — Nephronophthisis, familial juvenile; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients with nephronophthisis/renal associated ciliopathies (Other): Affected patients:
  Suffering from nephronophthisis or renal associated ciliopathies with known genetic diagnosis or not, Having obtained the signature of the informed consent form of patient, parent
  Intervention : blood and urine sample collection Collection of urines from patients will be followed by multiomics analyses including proteome and miRNAome profiling on EVs purified from urines by ultracentrifugation and metabolomics on unfractionated urine. Biomarkers identification for ciliopathy-induced chronic kidney disease will allow to monitor the drug response in treated urine-derived renal epithelial cells.
  Interventions: Other: Description: Research of therapeutic targets in the frame of nephronophthisis and renal associated ciliopathie
- Healthy relatives of Patients (Other): Healthy relatives:
  Being the healthy relative (father / mother / brother / sister) of an included patient Having signed the informed consent form (patient or parent in case of minor subject) No age limit is requested for these subjects, who can be recruited from birth.
  Intervention : blood and urine sample collection Collection of urines from patients will be followed by multiomics analyses including proteome and miRNAome profiling on EVs purified from urines by ultracentrifugation and metabolomics on unfractionated urine. Biomarkers identification for ciliopathy-induced chronic kidney disease will allow to monitor the drug response in treated urine-derived renal epithelial cells
  Interventions: Other: Description: Research of therapeutic targets in the frame of nephronophthisis and renal associated ciliopathie
- Negative control (Other): Being unscathed of any chronic renal disease, with or without ciliopathies Having obtained the signature of the informed consent form No age limit is requested for these patients, who can be recruited from birth.
  Intervention : blood and urine sample collection Collection of urines from patients will be followed by multiomics analyses including proteome and miRNAome profiling on EVs purified from urines by ultracentrifugation and metabolomics on unfractionated urine. Biomarkers identification for ciliopathy-induced chronic kidney disease will allow to monitor the drug response in treated urine-derived renal epithelial cells
  Interventions: Other: Description: Research of therapeutic targets in the frame of nephronophthisis and renal associated ciliopathie
- Positive control (Other): Suffering from Chronic Kidney Disease unrelated to ciliary dysfunction (such as glomerulopathy, tubulopathy…) Having obtained the signature of the informed consent form No age limit is requested for these patients, who can be recruited from birth.
  Intervention : blood and urine sample collection Collection of urines from patients will be followed by multiomics analyses including proteome and miRNAome profiling on EVs purified from urines by ultracentrifugation and metabolomics on unfractionated urine. Biomarkers identification for ciliopathy-induced chronic kidney disease will allow to monitor the drug response in treated urine-derived renal epithelial cells
  Interventions: Other: Description: Research of therapeutic targets in the frame of nephronophthisis and renal associated ciliopathie

INTERVENTIONS:
Other: Description: Research of therapeutic targets in the frame of nephronophthisis and renal associated ciliopathie

SUMMARY:
Nephronophthisis (NPH) is an autosomal recessive, genetically heterogeneous disease, with mutations identified in over 20 genes (notably NPHP1 and NPHP4).

These genetic defects are associated with reduced urine concentration, chronic tubulointerstitial nephritis, etc., and progress to end-stage renal failure before the age of 20.

Nephronophthisis may occur as an isolated pathology, but is also often associated with various extrarenal symptoms.

NPHP genes account for around 50% of the genes responsible for NPH. No effective treatment is available to date.

Studying NPHP proteins and associated signaling pathways could help identify how to circumvent the problems of protein distribution and therapeutic mRNA, and could be applicable to a broad set of NPHP mutations. To this end, Dr. Saunier's laboratory at Institut Imagine has recently identified approved drugs that correct some of the ciliary and epithelial defects found in cells with NPHP mutations.

DETAILED DESCRIPTION:
Nephronophthisis (NPH) is an autosomal recessive, genetically heterogeneous disease, with mutations identified in over 20 genes (notably NPHP1 and NPHP4).

These genetic defects are associated with reduced urine concentration, chronic tubulointerstitial nephritis, etc., and progress to end-stage renal failure before the age of 20.

Nephronophthisis may occur as an isolated pathology, but is also often associated with various extrarenal symptoms such as retinal dystrophy, cerebellar vermis hypoplasia, skeletal dysmorphisms and/or situs/inversus. These disorders overlap phenotypically, genetically and functionally. All are thought to result from defective ciliary signaling and are classified as renal ciliopathies.

NPHP genes account for around 50% of the genes responsible for NPH. No effective treatment is available to date.

One possible therapeutic approach is to replace the defective protein; but delivery of recombinant proteins or mRNA to renal tubular cells is not currently feasible. However, each NPHP protein participates in numerous intracellular signalling pathways involving cilia functions.

Studying NPHP proteins and associated signaling pathways could help identify how to circumvent the problems of protein distribution and therapeutic mRNA, and could be applicable to a broad set of NPHP mutations. To this end, Dr. Saunier's laboratory at Institut Imagine has recently identified approved drugs that correct some of the ciliary and epithelial defects found in cells with NPHP mutations.

The global research project of which this protocol is a part seeks to identify new specific targets and develop new therapeutic agents against these targets for the treatment of NPH and other ciliopathies.

ELIGIBILITY:
Inclusion Criteria:

* In order to be included in the protocol, subjects will have to respect the following criteria:

Affected patients:

Suffering from nephronophthisis or renal associated ciliopathies with known genetic diagnosis or not, Having obtained the signature of the informed consent form of patient, parent(s) or legal representative No age limit is requested for these patients, who can be recruited from birth.

Healthy relatives:

Being the healthy relative (father / mother / brother / sister) of an included patient Having signed the informed consent form (patient or parent in case of minor subject) No age limit is requested for these subjects, who can be recruited from birth.

'Negative' control patients: Being unscathed of any chronic renal disease, with or without ciliopathies Having obtained the signature of the informed consent form No age limit is requested for these patients, who can be recruited from birth.

'Positive' control patients Suffering from Chronic Kidney Disease unrelated to ciliary dysfunction (such as glomerulopathy, tubulopathy…) Having obtained the signature of the informed consent form No age limit is requested for these patients, who can be recruited from birth.

Exclusion Criteria:

In order to be included in the protocol, subjects will have to fulfill none of the following criteria:

Affected patients:

Patients with a functioning kidney transplant (only for patient for who urine sample is performed. This criteria is not applicable when only blood is sampling) Patients included in a therapeutic protocol since fewer 30 days.

Healthy relatives:

No no-inclusion criteria

'Negative' control subjects: No no-inclusion criteria

'Positive' control subjects: Patients with a functioning kidney transplant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Positive or negative confirmation of potential therapeutic targets in urine-derived renal epithelial cells of patients | 3 years

SECONDARY OUTCOMES:
Experimental transcriptomics data package from in vitro tubule cell model perturbed with disease network modifying agents | 3 years
  The experimental design and data will be formatted for Bayesian analytics.
A rank ordered list of specific druggable nodes within the NPHP disease module that could be targeted by biologic or chemical entities. | 3 years
  A rank ordered list of specific druggable nodes within the NPHP disease module that could be targeted by biologic or chemical entities.
Identify biomarkers to evaluate the response to small molecules for the management of NPHP and other renal ciliopathies. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Imagine Institute, La Defense, France

IPD SHARING:
Plan to Share IPD: Undecided